CLINICAL TRIAL: NCT03087240
Title: Influence of Dental Prophylaxis on Disease Activity of Rheumatoid Arthritis
Brief Title: Dental Prophylaxis and Rheumatoid Arthritis
Acronym: PREPARA II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Diana Wolff, Deputy Medical Director, Department of Conservative Dentistry, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: S-130/2016
Record Dates: First submitted 2017-03-15; First posted 2017-03-22 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis; Periodontitis; Gingivitis; Dental Prophylaxis
Keywords: Disease Activity Score 28 (DAS28); Health Assessment Questionnaire (HAQ); Dental Scaling; Dental Polishing; Oral Health; Gingival Crevicular Fluid; Inflammatory Cytokine Profile; Biofilm; Oral Microbiome; Intestinal Microbiome
MeSH Terms: conditions — Arthritis, Rheumatoid; Periodontitis; Gingivitis | interventions — Dental Prophylaxis; Dental Scaling; Dental Polishing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Dental Prophylaxis at fist visit (T0), after 2 weeks (T1) and after 3 months (T2)
  Interventions: Procedure: Dental Prophylaxis
- Control (Other): Wait & Control Study Design: Dental Prophylaxis after 3 months (T2) only
  Interventions: Procedure: Dental Prophylaxis

INTERVENTIONS:
Procedure: Dental Prophylaxis — Prevention and treatment of periodontal diseases by cleaning of the teeth in the dental office using the procedures of dental scaling and dental polishing. The treatment includes plaque detection, removal of supra- and subgingival plaque and calculus, as well as motivation and demonstration for establishing a sufficient oral hygiene.
  Other Names: Professional Teeth Cleaning; Dental Scaling; Dental Polishing

SUMMARY:
This study evaluates the influence of dental prophylaxis on disease activity of Rheumatoid Arthritis. In addition to standard antirheumatic therapy, recently the question has been raised whether or not there is a supplementary beneficial effect due to professional teeth cleaning. So far just a few studies pursued this question, indicating that prophylaxis by dental professionals can alleviate the symptoms of Rheumatoid Arthritis. To further evaluate this question, in our study half of the participants will receive dental prophylaxis at their first visit, after 2 weeks and 3 months, while the other half will receive professional teeth cleaning after 3 months only.

DETAILED DESCRIPTION:
Periodontitis (PA) and Rheumatoid Arthritis (RA) both rely on an over-regulated immune response, leading to inflammation in joints and periodontium. It is known, that both diseases have a reciprocal influence and that therapy of one disease may have beneficial effects on the course of the other.

This study evaluates the influence of dental prophylaxis on disease activity of Rheumatoid Arthritis, in addition to standard antirheumatic therapy. Patients are being recruited from the Department of Rheumatology at the Heidelberg University Hospital. Patients being diagnosed with an active Rheumatoid Arthritis (DAS28-Score > 3.2) will be included into the current study.

The study follows a prospective, randomized, controlled study design with the participating dental and rheumatologic investigators being both blinded. The first visit (T0) includes the assessment of demographic and disease-related parameters, such as quality of life (HAQ - Health Assessment Questionnaire) and disease activity (DAS28 - Disease Activity Score 28) by a rheumatologist. Afterwards a dental investigator will determine the status of oral health with standard parameters (periodontal status (pocket depth, attachment level, Bleeding on Probing (BPI)) and dental status (DMFT - Decayed Missing Filled Teeth)). Subsequently patients are being randomized 1:1. The dental intervention is defined as a standardized dental prophylaxis according to the Heidelberg Therapeutic Scheme for Hygienization of the Oral Condition by means of professional teeth cleaning and motivational and demonstrational measures for implementing a sufficient oral hygiene.

Group 1 (Test) contains patients being randomized for the dental intervention at first visit. Accordingly Group 2 (Control) contains patients not being randomized for the dental intervention. After 14 days (T1) patients in Group 1 undergo once again dental prophylaxis according the Heidelberg Therapeutic Scheme. The next follow-up is being executed after 3 months (T2) by rheumatologic and dental investigators again. The primary outcome consists of the evaluation of the disease activity of the Rheumatoid Arthritis measured by the DAS28-Score between first visit (T0) and after 3 months (T2). Patients of Group 2 receive dental prophylaxis after 3 months due to ethical reasons ("Wait & Control Study Design"). The final visit takes place after an additional 3 months (T3), in order to evaluate a possible long-term effect of the dental intervention.

Furthermore the development of the bacterial microflora and inflammatory cytokine profile is being investigated. For this purpose, samples of supra- and subgingival plaque, gingival crevicular fluid and saliva at visits T0, T2 and T3 as well as stool samples at T0 and T2 are being collected. These will be analyzed qualitatively and quantitatively by molecular genetic methods.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form
* Diagnosis of an active Rheumatoid Arthritis (DAS28 > 3.2) by a rheumatologist
* Gingiva Bleeding Index (GBI) > 10%, Plaque Control Record (PCR) > 30% (indication for Dental Prophylaxis following the Heidelberg Therapeutic Scheme)

Exclusion Criteria:

* Generalized Severe Chronic Periodontitis
* Periodontal treatment within the last 6 months
* Dental Prophylaxis within the last 6 months
* Dental Prophylaxis being contraindicated due to dental or other reasons
* Antibiotic treatment within the last 3 months (excluding intake of antibiotic prophylaxis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Disease Activity Score 28 (DAS28) | baseline (T0) and three months (T2)
  The Disease Activity Score 28 (DAS28) combines single measures into an overall, continuous measure of Rheumatoid Arthritis disease activity. The DAS28 includes a 28 tender joint count, a 28 swollen joint count, acute phase reactant and a general health assessment on a visual analog scale.

SECONDARY OUTCOMES:
Health Assessment Questionnaire (HAQ) | baseline (T0) and three months (T2)
  The Health Assessment Questionnaire (HAQ) is a comprehensive, validated, patient-oriented outcome assessment instrument. It includes the five dimensions disability, pain, medication effects, costs of care and mortality, which are then further subcategorized.
Microbiome and Inflammatory Cytokine Profile | baseline (T0), three months (T2) and six months (T3)
  The development of the bacterial microflora and inflammatory cytokine profile is being analyzed qualitatively and quantitatively by molecular genetic methods. Samples of supra- and subgingival plaque, gingival crevicular fluid and saliva are being collected at T0, T2 and T3, stool samples are being collected at T0 and T2.
Cumulative Steroid Dose | baseline (T0), three months (T2) and six months (T3)
  The cumulative steroid dose is being compared between Group 1 (Test) and Group 2 (Control).

CONTACTS AND LOCATIONS:
Overall Officials: Diana Wolff, Prof. Dr. med. dent., Principal Investigator — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janssen KM, Vissink A, de Smit MJ, Westra J, Brouwer E. Lessons to be learned from periodontitis. Curr Opin Rheumatol. 2013 Mar;25(2):241-7. doi: 10.1097/BOR.0b013e32835d833d. PMID 23370377
- [Background] Ortiz P, Bissada NF, Palomo L, Han YW, Al-Zahrani MS, Panneerselvam A, Askari A. Periodontal therapy reduces the severity of active rheumatoid arthritis in patients treated with or without tumor necrosis factor inhibitors. J Periodontol. 2009 Apr;80(4):535-40. doi: 10.1902/jop.2009.080447. PMID 19335072